CLINICAL TRIAL: NCT06802367
Title: Environmental Exposures in a Clinical Setting: the Impact on Patients
Brief Title: Hospital Environmental Exposure
Status: Not yet recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0988
Record Dates: First submitted 2024-12-10; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Environment; Sleep; Noise Exposure; Air Quality; Light
Keywords: Air quality; Noise; Light; Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Environmental data collected (noise, light and air quality levels). Body temperature, heart rate and measurements of patient sleep using wearable sensors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is an increasing body of evidence that human health is affected by environmental factors such as air quality, noise and light. This applies to both indoor and outdoor environments. While there have been several studies looking at homes, offices and work environments, hospital environments are still poorly characterised. Indoor hospital environments are complex, and patients with various health conditions can spend extended periods of time in wards. A number of studies have reported an association of air pollution exposure and a disturbance to sleep. A lack of sleep, or poor and disrupted sleep can impact health. Disturbed sleep therefore can impact a patient's recovery in hospital wards. In addition to the exposure to air pollutants, noise and light levels within the hospital environment can also have an impact on patient health. Inadequate, or a disrupted light and dark cycles can impact the circadian rhythm of the human body, responsible for the sleep cycle. In this study, the investigators aim to characterise these exposures and address the impact of these exposures on the patient sleep. Given the links between sleep and the environmental conditions.

DETAILED DESCRIPTION:
The proposed study will aim to answer the research question- Can a method be developed to assess the impact of environmental exposures on patient sleep in a clinical setting?

There are very few health-based guidelines regarding hospital indoor environments. With regards to noise in hospital wards, the World Health Organisation (WHO) have recommended that noise in hospital wards should not exceed 30 dB at night, however owing to excessive noise generated by a number of factors, these noise levels can be larger, up to 75 dB within intensive care units and 45 dB in emergency departments. Noise therefore is a common complaint from patients with regards to disrupting their sleep. There are also no clear guidelines on light levels in clinical settings. The link between sleep and health is well known. Sleep is not just a period of inactivity or unconsciousness but is a complex physiological process composed of repeated cycles of non-rapid eye movement (NREM) and rapid eye movement (REM). A lack of, or poor sleep can disturb a patients circadian rhythm, changing body temperature (where core temperature changes with sleep- wake cycles), and changing heart rate. In a hospital ward, there are a number of environmental factors that can disturb a patient's sleep. It is therefore important to assess the contributors to poor sleep in a clinical environment and mitigate the adverse effects of poor air quality, light and noise to improve patient sleep. The aim with this work is therefore two-fold. The investigators aim to collect pilot data that quantitatively characterises the indoor environment within a clinical setting in terms of air quality, noise and light. The approach will use, sound level meters, air quality sensors and light level meters installed within a hospital ward to characterise the hospital environment that patients experience. Such techniques provide a meaningful description of the clinical environmental conditions. The data collected will be compared against any available health guidelines. A further aim to assess the impact of these environmental conditions on patient sleep as adequate sleep is essential to health.

To assess the patients, the investigators will be using actigraphy (accelerometer worn on the wrist or arm) activity monitors for sleep monitoring. The participant will also be given a second wearable monitor that will measure their heart rate and body temperature. The data collected from the two wearable monitors will be compared with environmental monitoring data (air quality, light and noise) in order to determine if environmental conditions are linked to sleep patterns. Sleep times, sleep efficiency, number of awakenings and sleep latency will be recorded from the sleep data. The participant will also be given a sleep diary will be used in order to assess the perceived quality of sleep. The sleep diary will be completed during the participants time in the ward and will ask the participant to note, sleep and awake times as well as any sources of disturbing light and noise within the ward in the participants opinion.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission with a diagnosis that requires at least 2 nights.
* Participant is willing and able to give informed consent for participation in the study. If a patient for example has dementia and/ or the inability to retain information or if they are unable to wear the device, they will not be consented.
* Aged 18 years or above.
* Able (in the ward staff, research team and investigator's opinion) and willing to comply with all study requirements.

Exclusion Criteria:

* Any significant disease or disorder which, in the opinion of the investigator, may either put the participants or other patients at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Reported history of sleep disorders, including obstructive sleep apnoea syndrome (OSAS) or insomnia.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: University Hospitals Leicester Patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Concentrations of nitrogen dioxide (NO2) in selected hospital wards | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Using air quality sensors installed within selected wards, the concentrations of NO2 (ugm-3) will be measured. Hourly averaged NO2 concentration data will be collected continuously until the end of the data collection period.
Comparisons of NO2 concentrations measured in selected hospital wards with published guidelines | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Concentrations of NO2 measured within wards will be compared with World Health Organisation (WHO) daily averaged and annual guidelines of NO2 concentrations. Measurements of NO2 will also be compared against UK hourly and annual mean guideline NO2 concentrations.
Concentrations of ozone (O3) in selected hospital wards | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Using air quality sensors installed within selected wards, the concentrations of O3 (ugm-3). Hourly averaged O3 concentration data will be collected continuously until the end of the data collection period.
Concentrations of particulate matter (PM2.5) in selected hospital wards | Through study completion, an average of 1 year, 11 months
  Using air quality sensors installed within selected wards, the concentrations of PM2.5 (ugm-3). Hourly averaged PM2.5 concentration data will be collected continuously until the end of the data collection period.
Comparisons of PM2.5 concentrations measured in selected hospital wards with published guidelines | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Concentrations of PM2.5 measured within wards will be compared with World Health Organisation (WHO) daily averaged and annual guidelines of PM2.5 concentrations. Measurements of PM2.5 will also be compared against UK guidelines of annual average PM2.5 concentrations.
Measurements of noise volume in selected hospital wards | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Portable noise monitors will be installed in selected hospital wards. The noise monitors will measure the volume of noise in wards in decibels (dB) continuously until the end of the data collection period.
Comparisons of measured volume in selected hospital wards with published guidelines | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  WHO have published guidelines of noise levels (in decibels) in hospitals at night and during the day. The measurements of noise collected in this study will be compared with WHO published guidelines.
Measurements of noise frequency in selected hospital wards | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Portable noise monitors will be installed in selected hospital wards. The noise monitors will measure the frequency of noise in wards (Hz).
The temperature in selected hospital wards will be measured. | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Using the air quality sensor installed within the ward, the temperature in degrees Celsius (°C) will be measured continuously.
Light illuminance measured in selected wards | From the start of the data collection period to June 2026, an average of 1 year, 6 months
  Portable light level meters will be installed in wards. Illuminance in lux (lx) will be measured continuously.
Total sleep time | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Measured using actigraphy, total sleep time will be measured (in hours). Measurements will be averaged per day and averaged over the total time the participant was included in the study.
Sleep Onset Latency | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  The time it takes a person to fall asleep after turning the lights off (measured in hours). Measured using actigraphy. Will be averaged per day and averaged over the total time the participant was included in the study.
Sleep Efficiency (%) | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Sleep Efficiency (%) = (Total Sleep Time (hours)/ Time in Bed (hours)) x 100 Measured using actigraphy. Will be averaged per day and averaged over the total time the participant was included in the study.
Wake after sleep onset | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Periods of wakefulness after a defined sleep onset. Calculated by the total time of the periods that are inside a sleep period but are not a sleep state (ex.: rest, awake) Measured using actigraphy. Measured in minutes. Will be averaged per day and averaged over the total time the participant was included in the study.
Number of awakenings | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  The number of rest/ awake periods. Measured using actigraphy. Will be averaged per day and averaged over the total time the participant was included in the study.
Number of naps | Up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Measured using actigraphy. Will be averaged per day and averaged over the total time the participant was included in the study.
Score on a Sleep Diary | Every morning for up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Participants will be asked to complete a sleep diary. The sleep diary will ask the participant to score their:
  Mood during the day (1 = lowest mood, 10= excellent mood), Tiredness during the day (1 = least tired, 10= most tired), Activity during the day? (1= least active, 10 = most active), Quality of your sleep in hospital? (1= worst, 10= excellent), On waking up in the morning, how rested do they feel? (1= least rested, 10= most rested), How disruptive was the noise in the ward to their sleep? (1= least disruptive, 10= most disruptive), How disruptive was the light in the ward to their sleep? (1 least disruptive, 10= most disruptive).
  This question will be asked every morning for 7 days. These questions will be asked every morning for 7 days.
Sleep Diary | Every morning for up to 7 days from the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Participants will be asked to complete a sleep diary. The sleep diary will ask the participant:
  How many naps did they take during the day? How long for? Time they went to sleep for the night Number of times they woke up in the night Number of hours they slept last night This question will be asked every morning for 7 days. This question will be asked every morning for 7 days.
Sleep Diary | From the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Participants will be asked to complete a sleep diary. The sleep diary will ask the participant, yes/ no questions on:
  Have you/are you currently using an eye mask in hospital? Have you/are you currently using an ear plugs in hospital? These questions will only be asked once
Score on a Sleep Diary | From the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Participants will be asked to complete a sleep diary. The sleep diary will ask the participant list and to score any disruptive noises within the hospital ward that impacts their sleep (1 is no disruption and 10 is significant disruption). This question will be asked once.
Sleep Diary- sleep at home | From the date of recruitment or until the participant moves ward or is discharged (whichever is first)
  Participants will be asked to complete a sleep diary. The sleep diary will also ask questions regarding their sleep at home:
  What time do you usually go to sleep at home? What time do you usually wake up in the mornings at home? On average, at home, how many hours a night do you usually sleep? Rate the quality of your usual sleep at home. (1= worst, 10= excellent). Yes/ No questions will also be asked regarding the participant wearing an eye mask and ear plugs at home.
  Space is also provided for the participant to add additional notes These questions will be asked once.

SECONDARY OUTCOMES:
Suggested interventions which could be used to improve the patient's environment within the hospital. | Through study completion, an average of 1 year, 11 months
  The patient will be asked to complete a sleep diary. The sleep diary will also ask the patient to list any environmental conditions (light or noise) that disturbs their sleep. This data will be used to suggest methods that can be used to improve the light and noise levels within that specific ward.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Vande Hey, PhD, Study Chair — University of Leicester; Antonella Ghezzi, Principal Investigator — University Hospitals, Leicester

REFERENCES:
- [Background] Fonseca A, Abreu I, Guerreiro MJ, Barros N. Indoor Air Quality in Healthcare Units- A Systematic Literature Review Focusing Recent Research. Sustainability. 2022;14(2)
- [Background] Berglund B, Lindvall T, Schwela DH. New WHO guidelines for community noise. Noise & Vibration Worldwide. 2000;31(4):24-29
- [Background] Emar M, Smith E, Coats TJ. Background noise in an Emergency Department: an observational study from staff and patient perspectives. medRxiv. 2022:2022.2005.2020.22275148
- [Background] Hillman DR. Sleep Loss in the Hospitalized Patient and Its Influence on Recovery From Illness and Operation. Anesth Analg. 2021 May 1;132(5):1314-1320. doi: 10.1213/ANE.0000000000005323. PMID 33857973
- [Background] Luyster FS, Strollo PJ Jr, Zee PC, Walsh JK; Boards of Directors of the American Academy of Sleep Medicine and the Sleep Research Society. Sleep: a health imperative. Sleep. 2012 Jun 1;35(6):727-34. doi: 10.5665/sleep.1846. PMID 22654183
- [Background] Lucchini A, Giani M, Ferrari K, Di Maria S, Galimberti G, Zorz A, Iozzo P, Elli S, Fumagalli R, Bambi S. Sound and Light Levels in a General Intensive Care Unit Without Windows to Provide Natural Light. Dimens Crit Care Nurs. 2023 Mar-Apr 01;42(2):115-123. doi: 10.1097/DCC.0000000000000569. PMID 36720036
- [Background] Xie H, Kang J, Mills GH. Clinical review: The impact of noise on patients' sleep and the effectiveness of noise reduction strategies in intensive care units. Crit Care. 2009;13(2):208. doi: 10.1186/cc7154. Epub 2009 Mar 9. PMID 19344486
- [Background] Touitou Y, Reinberg A, Touitou D. Association between light at night, melatonin secretion, sleep deprivation, and the internal clock: Health impacts and mechanisms of circadian disruption. Life Sci. 2017 Mar 15;173:94-106. doi: 10.1016/j.lfs.2017.02.008. Epub 2017 Feb 16. PMID 28214594
- [Background] Boivin DB, Duffy JF, Kronauer RE, Czeisler CA. Dose-response relationships for resetting of human circadian clock by light. Nature. 1996 Feb 8;379(6565):540-2. doi: 10.1038/379540a0. PMID 8596632
- [Background] Elbaz M, Leger D, Sauvet F, Champigneulle B, Rio S, Strauss M, Chennaoui M, Guilleminault C, Mira JP. Sound level intensity severely disrupts sleep in ventilated ICU patients throughout a 24-h period: a preliminary 24-h study of sleep stages and associated sound levels. Ann Intensive Care. 2017 Dec;7(1):25. doi: 10.1186/s13613-017-0248-7. Epub 2017 Mar 3. PMID 28255956
- [Background] Sanchez T, Gozal D, Smith DL, Foncea C, Betancur C, Brockmann PE. Association between air pollution and sleep disordered breathing in children. Pediatr Pulmonol. 2019 May;54(5):544-550. doi: 10.1002/ppul.24256. Epub 2019 Feb 4. PMID 30719878
- [Background] Tsai LJ, Yuan TH, Shie RH, Chiang CH, Chan CC. Association between ambient air pollution exposure and insomnia among adults in Taipei City. Sci Rep. 2022 Nov 9;12(1):19064. doi: 10.1038/s41598-022-21964-0. PMID 36351973
- [Background] Oliveira L, Gomes C, Bacelar Nicolau L, Ferreira L, Ferreira R. Environment in pediatric wards: light, sound, and temperature. Sleep Med. 2015 Sep;16(9):1041-8. doi: 10.1016/j.sleep.2015.03.015. Epub 2015 Apr 27. PMID 26298777
- [Background] Cincinelli A, Martellini T. Indoor Air Quality and Health. Int J Environ Res Public Health. 2017 Oct 25;14(11):1286. doi: 10.3390/ijerph14111286. PMID 29068361
- [Background] Stansfeld SA, Matheson MP. Noise pollution: non-auditory effects on health. Br Med Bull. 2003;68:243-57. doi: 10.1093/bmb/ldg033. PMID 14757721
- [Background] GBD 2017 Risk Factor Collaborators. Global, regional, and national comparative risk assessment of 84 behavioural, environmental and occupational, and metabolic risks or clusters of risks for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1923-1994. doi: 10.1016/S0140-6736(18)32225-6. Epub 2018 Nov 8. PMID 30496105